CLINICAL TRIAL: NCT03707028
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Rivoceranib in Combination With Paclitaxel in Advanced Gastric or Gastroesophageal Junction Cancer
Brief Title: A Study to Evaluate Safety, Tolerability, and Efficacy Profile of Rivoceranib With Paclitaxel in Advanced Gastric or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated after completion of Part 1 due to a change in research plan.
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSK-RM109
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rivoceranib with Paclitaxel (Experimental): Participants will receive oral daily doses of rivoceranib per 28-day cycle (as its mesylate salt) with a fixed dose of paclitaxel given intravenously on Day 1, Day 8, and Day 15 of the 28-day cycle.
  Interventions: Drug: Rivoceranib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Rivoceranib — Film-coated tablet
  Other Names: Apatinib
Drug: Paclitaxel — Solution administered intravenously
  Other Names: Taxol

SUMMARY:
This is an open-label, single-center, single-arm, dose escalation and dose expansion Phase I/IIa study designed to determine the recommended Phase 2 dose (RP2D) and the safety and tolerability profile along with preliminary signs of efficacy of rivoceranib in combination with paclitaxel as a second-line therapy in advanced, recurrent and/or metastatic gastric or gastroesophageal junction cancer. This study will also characterize the pharmacokinetic (PK) parameters of rivoceranib and paclitaxel when given in combination.

DETAILED DESCRIPTION:
Primary Phase I Objectives

* To determine the RP2D dose of rivoceranib in combination with paclitaxel.

Primary Phase II Objectives

* To determine clinical activity of the combination of rivoceranib and paclitaxel.

Secondary Phase I Objectives

* To evaluate the PK of rivoceranib and paclitaxel when given in combination.
* To assess the efficacy of rivoceranib in combination with paclitaxel.

Secondary Phase II Objectives

* To assess the efficacy of rivoceranib in combination with paclitaxel.
* To assess the safety and tolerability of rivoceranib in combination with paclitaxel.
* To assess the PK of rivoceranib and paclitaxel when given in combination.

ELIGIBILITY:
Inclusion Criteria

1. Participants with documented locally advanced unresectable or metastatic gastric or gastroesophageal junction cancer refractory to or relapsing after first line platinum and fluoropyrimidine containing chemotherapy (with or without trastuzumab) with an indication for therapy with paclitaxel and an antiangiogenic agent. If disease progression occurs during or within 6 months after completion of any adjuvant chemotherapy, this therapy is considered a first-line chemotherapy for participant eligibility.
2. Participants who have provided tumor tissue prior to initiation of first-line therapy and have provided or can provide tumor tissue prior to screening in this study. This will be optional for Phase I participants. Tumor tissue must not have been irradiated.
3. Participants who have at least 1 measurable lesion as defined by RECIST v1.1. This will be optional for Phase I participants.
4. Adequate bone marrow, renal, and liver function evidenced by:

   1. Hematologic: Absolute neutrophil count of ≥1,500/cubic millimeter (mm^3), platelet count of ≥ 1,00,000/mm ^3, and hemoglobin of ≥9.0 grams (g)/deciliter (dL). Transfusion of platelets or red blood cells to meet the inclusion criteria within 2 weeks of screening is not allowed.
   2. Adequate renal function, defined as meeting any 1 of the following criteria:

   i. Serum creatinine <1.5 × upper limit of normal (ULN). ii. Creatinine clearance based on the Cockcroft-Gault estimate ≥50 milliliters per minute (mL/min) or creatinine clearance based on urine collection (12 or 24 hours) ≥50 mL/min.

   iii. In addition, urinary protein should be <2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24 hour urine or urine protein/creatinine ratio must be collected and must demonstrate <2 g of protein in 24 hours.

   c) Hepatic: Serum bilirubin <1.5 × ULN, aspartate and alanine aminotransferase ≤3.0 × ULN (≤5.0 × UNL, if with liver metastases). If liver and/or bone metastases alkaline phosphatase ≤5 × ULN.
5. Blood coagulation tests: Prothrombin time and international normalized ratio ≤1.5 × ULN.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Estimated life expectancy of at least 12 weeks.
8. Ability to swallow the study drug without chewing, breaking, crushing, opening or otherwise altering the product formulation. If vomiting occurs, the dose will not be replaced. Antiemetics must be used at efficacious doses.
9. No major gastrointestinal disease (e.g., chronic diarrheal disease) or intestinal surgery that can jeopardize drug absorption.

Exclusion Criteria

1. Prior use of taxane (paclitaxel or docetaxel) or any contraindication for therapy with paclitaxel.
2. Previous treatment with rivoceranib or any other systemic therapy with a vascular endothelial growth factor (VEGF) pathway inhibitor.
3. Known hypersensitivity to rivoceranib or any component of its formulation or history of severe adverse events, including uncontrolled hypertension or other common anti-angiogenesis drug class effects during prior exposure to vascular inhibitors.
4. Any unresolved toxicity Grade >1 (except alopecia) from previous anticancer therapy (including radiotherapy).
5. Has history of another malignancy within 2 years prior to screening. Participants with the following are eligible for this study if, in the opinion of the investigator, they do not pose a significant risk to life expectancy:

   1. Bladder tumors considered superficial such as noninvasive (T1a) and carcinoma in situ (Tis).
   2. Curatively treated cervical carcinoma in situ.
   3. Thyroid papillary cancer with prior treatment.
   4. Carcinoma of the skin without melanomatous features.
   5. Prostate cancer which has been surgically or medically treated and not likely to recur within 2 years.
6. Known brain metastasis or other central nervous system metastasis that is either symptomatic or untreated. Metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by computed tomographic scan at least 4 weeks before screening without evidence of cerebral edema. Participants on stable dose of corticosteroids or anticonvulsants are permitted.
7. Has received prior anticancer therapy within 3 weeks before Cycle 1 Day 1. Traditional herbal remedies with anti-infective, immune stimulating, or anticancer properties are not allowed from screening throughout the entire period of study participation.
8. Current or recent (within 10 days of Cycle 1 Day 1) use of full dose oral or parenteral anticoagulants or other thrombolytic agents for therapeutic (as opposed to prophylactic) purposes, clinically serious non-healing wounds, or incompletely healed bone fracture. A maximum dose of 325 milligrams (mg)/day of aspirin is allowed.
9. Participants who had therapeutic paracentesis of ascites (>1 liter [L]) within the 2 months prior to starting study treatment or who, in the opinion of the investigator, will likely need therapeutic paracentesis of ascites (>1L) within 2 months of Cycle 1 Day 1.
10. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9, and CYP2C19.
11. Active bacterial infections (including tuberculosis and syphilis) requiring systemic antibiotic therapy.
12. Known history of human immunodeficiency virus infection.
13. Active hepatitis B or C infection or chronic hepatitis B or C infection requiring treatment with antiviral therapy or prophylactic antiviral therapy; unless evidence of viral suppression has been documented and the participant will remain on appropriate antiviral therapy throughout the study.
14. Child-Pugh Stage B and C liver function impairment.
15. Pregnant or breastfeeding women. Participants unwilling to comply with birth control requirements will not be eligible.
16. History of uncontrolled hypertension (blood pressure ≥140/90 mmHg and change in antihypertensive medication within 7 days prior to screening) that is not well managed by medication and the risk of which may be precipitated by a VEGF inhibitor therapy. History of hypertensive crisis, and hypertensive encephalopathy.
17. Participants who have a known history of symptomatic congestive heart failure (New York Heart Association III to IV), symptomatic or poorly controlled cardiac arrhythmia, complete left bundle branch block, bifascicular block, or any clinically significant ST segment and/or T wave abnormalities, corrected QT interval by Fredericia (QTcF) > 450 msec for males or QTcF > 470 milliseconds (msec) for females prior to screening.
18. History of bleeding diathesis or clinically significant bleeding within 14 days prior to Cycle 1 Day 1. This includes a history of gastrointestinal bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3 months prior to Cycle 1 Day 1 that, in the investigator's opinion, may place the participant at risk of side effects from anti-angiogenesis products.
19. History of clinically significant thrombosis (bleeding or clotting disorder) within the past 3 months prior to Cycle 1 Day 1 that, in the investigator's opinion, may place the participant at risk of side effects from anti-angiogenesis products.
20. History of other significant cardiovascular diseases or vascular diseases within the last 6 months prior to screening (e.g., myocardial infarction or unstable angina pectoris, stroke or transient ischemic attack, or significant peripheral vascular diseases) that, in the investigator's opinion, may pose a risk to the participant on vascular endothelial growth factor receptors (VEGFR) inhibitor therapy.
21. History of clinically significant glomerulonephritis, biopsy-proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies.
22. Psychological, familial, sociological, or geographical conditions including drug or alcohol abuse that do not permit compliance with the study participation or evaluation of the study results.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of Dose-Limiting Toxicities (DLT) During Cycle 1 | Cycle 1 (first 28 days)
  The number and proportion of participants experiencing DLTs will be reported by dose level, based on DLT observations during Cycle 1. Each Cycle is 28 days.
Phase I: Number of Participants Reporting Adverse Events (AEs) and Serious AEs (SAEs) | Up to 24 months
  An AE is any untoward medical occurrence in a participant or participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, or important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent 1 of the other outcomes listed above.
Phase II: Objective Response Rate (ORR) | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  ORR is the percentage of participants who achieve objective tumor response (complete response [CR] or partial response [PR]) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria for response.

SECONDARY OUTCOMES:
Phase I: Maximum Observed Concentration (Cmax) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Time to Maximum Observed Concentration (tmax) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC0-t) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Terminal Half-life (t1/2) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Apparent Oral Plasma Clearance (CL/F) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Apparent Volume of Distribution (Vz/F) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: Terminal Rate Constant (λz) | Day 1 & 15 of Cycle 1 (each cycle is 28 days)
Phase I: ORR | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  ORR by RECIST 1.1
Phase I: Progression-free Survival (PFS) | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  Defined as time from first dose of study drug (Cycle 1 Day 1) to the time of first documented disease progression or death due to any cause.
Phase I: Overall survival (OS) | Ongoing assessment from enrollment until end of study, up to approximately 24 months
  OS is the time from first dose of study drug (Cycle 1 Day 1) to the time of death from any cause.
Phase I: Disease Control Rate (DCR) | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  DCR is defined as the percentage of participants who achieve CR or PR and stable disease (SD) at ≥12 weeks.
Phase I: Duration of Response | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  Defined as the time from first documentation of (complete response or partial response) to the first documentation of progression.
Phase II: PFS | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  Defined as time from first dose of study drug (Cycle 1 Day 1) to the time of first documented disease progression or death due to any cause.
Phase II: OS | Ongoing assessment from enrollment until end of study, up to approximately 24 months
  OS is the time from first dose of study drug (Cycle 1 Day 1) to the time of death from any cause.
Phase II: DCR | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  DCR is defined as the percentage of participants who achieve CR or PR and SD at ≥12 weeks.
Phase II: Duration of Response | Every other cycle (each cycle is 28 days) until end of study, assessed up to 24 months
  Defined as the time from first documentation of (complete response or partial response) to the first documentation of progression.
Phase II: Number of Participants With AEs and SAEs | Ongoing assessment from enrollment until end of study, approximately 24 months
  Adverse Events and Serious Adverse Events
Phase II: Concentration at the End of the Dosage Interval (Ctrough) | Ongoing assessment from enrollment until end of study, approximately 24 months
  Ctrough is characterized at steady state after single and multiple cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, Dr., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea